CLINICAL TRIAL: NCT03779789
Title: Assessing Tolerability and Efficacy of Vortioxetine Versus SSRIs in Elderly Patients With Depression: a Pragmatic, Multicenter, Open-label, Parallel-group, Superiority, Randomized Trial
Brief Title: Vortioxetine in the Elderly vs. Selective Serotonin Reuptake Inhibitors (SSRIs): a Pragmatic Assessment
Acronym: VESPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: University of Catania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-0234923; 2018-001444-66 (EudraCT Number)
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder
Keywords: vortioxetine; SSRI; depression; elderly
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vortioxetine; Sertraline; Citalopram; Escitalopram; Paroxetine; Fluoxetine; Fluvoxamine

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicenter, open-label, parallel-group, superiority, randomized trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine
- SSRIs (Active Comparator)
  Interventions: Drug: Sertraline; Drug: citalopram; Drug: Escitalopram; Drug: Paroxetine; Drug: Fluoxetine; Drug: Fluvoxamine

INTERVENTIONS:
Drug: Vortioxetine — Antidepressant classified under the category "other antidepressants" according to the ATC/DDD index [ATC=Anatomical Therapeutic Chemical Classification System; DDD=Defined Daily Dose]. The dose will be flexible according to the clinical evaluation and in accordance with doses reported for elderly in the Summaries of Product Characteristics (available: https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/home) (namely: 5-20 mg/day).
  Other Names: Brintellix; Trintellix
  Arms: vortioxetine
Drug: Sertraline — Antidepressant classified under the category "Selective serotonin reuptake inhibitors" according to the ATC/DDD index. The dose will be flexible according to the clinical evaluation and in accordance with doses reported for elderly in the Summaries of Product Characteristics (available: https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/home) (namely: 50-200 mg/day).
  Other Names: Zoloft
  Arms: SSRIs
Drug: citalopram — Antidepressant classified under the category "Selective serotonin reuptake inhibitors" according to the ATC/DDD index. The dose will be flexible according to the clinical evaluation and in accordance with doses reported for elderly in the Summaries of Product Characteristics (available: https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/home) (namely: 10-20 mg/day).
  Other Names: Elopram
  Arms: SSRIs
Drug: Escitalopram — Antidepressant classified under the category "Selective serotonin reuptake inhibitors" according to the ATC/DDD index. The dose will be flexible according to the clinical evaluation and in accordance with doses reported for elderly in the Summaries of Product Characteristics (available: https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/home) (namely: 5-10 mg/day).
  Other Names: Entact
  Arms: SSRIs
Drug: Paroxetine — Antidepressant classified under the category "Selective serotonin reuptake inhibitors" according to the ATC/DDD index. The dose will be flexible according to the clinical evaluation and in accordance with doses reported for elderly in the Summaries of Product Characteristics (available: https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/home) (namely: 20-40 mg/day).
  Other Names: Daparox
  Arms: SSRIs
Drug: Fluoxetine — Antidepressant classified under the category "Selective serotonin reuptake inhibitors" according to the ATC/DDD index. The dose will be flexible according to the clinical evaluation and in accordance with doses reported for elderly in the Summaries of Product Characteristics (available: https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/home) (namely: 20-60 mg/day).
  Other Names: Prozac
  Arms: SSRIs
Drug: Fluvoxamine — Antidepressant classified under the category "Selective serotonin reuptake inhibitors" according to the ATC/DDD index. The dose will be flexible according to the clinical evaluation and in accordance with doses reported for elderly in the Summaries of Product Characteristics (available: https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/home) (namely: 100-300 mg/day).
  Arms: SSRIs

SUMMARY:
Background. Depression is a highly frequent condition in the elderly, with a huge impact on quality of life, life expectancy, and medical outcomes. SSRIs are commonly prescribed in elderly depressed patients and, although generally safe, they may be associated with tolerability issues. Based on available studies, vortioxetine is likely to have a promising tolerability profile in the elderly, as it does not adversely affect psychomotor or cognitive performance, wakefulness, body weight, and electrocardiogram parameters.

Objectives. Assessing the comparative tolerability, safety and efficacy of vortioxetine compared with the SSRIs as a group (including sertraline, citalopram, escitalopram, paroxetine, fluoxetine, fluvoxamine) in elderly patients affected by major depression. The primary outcome will be the withdrawal rate due to adverse events.

Methods. This is a pragmatic, multicenter, open-label, parallel-group, superiority, randomized trial. Twelve Italian Community Psychiatric Services will consecutively enrol elderly patients suffering from an episode of major depression who get in contact over a period of 12 months. By employing the web-based application RedCap, doctors will be able to randomize patients to vortioxetine or one of the SSRIs, chosen on the basis of clinical judgment, and to collect basic socio-demographic and clinical data. Trained and blinded assessors will administer five validated rating scales: Montgomery-Åsberg Depression Rating Scale (MADRS), Antidepressant Side-Effect Checklist (ASEC), EuroQual 5 Dimensions (EQ-5D), Charlson Age-Comorbidity Index (CACI), and Short Blessed Test (SBT). Patients will be assessed after 1, 3 and 6 months.

Expected results. On the basis of current literature, the investigators hypothesize vortioxetine to be superior to SSRIs as a group in terms of tolerability. As vortioxetine is expected to reduce the withdrawal rates due to adverse events of about 12% compared to SSRIs, and assuming that about 23% of the participants could be lost within 6 months, the investigators aim to enrol 358 patients (179 in each group).

ELIGIBILITY:
Inclusion Criteria:

1. 65 years old or above;
2. willing to participate by signing an informed consent;
3. suffering from an episode of major depression, based on clinical judgment (guided by DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) criteria);
4. treatment with an antidepressant is clinically appropriate, based on clinical/medical judgment;
5. agreement between investigator and patient to discontinue any current antidepressant, second generation antipsychotic, or lithium. According to the pragmatic design of the study, the discontinuation will be performed according to common routine practice. No specific protocols for discontinuation will be applied. All other concomitant medications are allowed;
6. uncertainty about which trial treatment would be best for the participant.

Exclusion Criteria:

1. dementia, of any type and stage, as formally diagnosed by a specialist (geriatrician, neurologist, or others);
2. diagnosis of schizophrenia or bipolar disorder;
3. clinical conditions or treatments which contraindicate the use of oral vortioxetine or SSRIs, according to clinical/medical judgment (for example conditions or treatments at high risk of bleeding, convulsions, serotoninergic syndrome, hyponatraemia, etc.). All concomitant medications will be prescribed according to routine clinical practice, in compliance with the synthesis of the product characteristics (Riassunto delle Caratteristiche del Prodotto - RCP) registered in the databank of the AIFA (Agenzia Italiana del Farmaco) (available at https://farmaci.agenziafarmaco.gov.it/bancadatifarmaci/cerca-farmaco).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 362 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants withdrawing from treatment due to adverse events (tolerability) | 6 months
  Participants withdrawing from allocated treatment due to adverse events on the number of randomized patients.

SECONDARY OUTCOMES:
Number of participants withdrawing from treatment due to any cause (acceptability) | 6 months
  Participants withdrawing from allocated treatment due to any cause on the number of randomized patients
Overall mortality | 6 months
  The number of deaths on the number of randomized patients
Number of participants with at least one episode of self-harm | 6 months
  Number of participants with at least one episode of self-harm on the number of randomized patients
Number of participants died by suicide | 6 months
  Number of participants died by suicide on the number of randomized patients
Treatment-related adverse events as assessed by the ASEC | 6 months
  The mean change score at the Antidepressant Side-Effect Checklist (ASEC). ASEC is a validated rating scale, administered by the clinician, measuring the occurrence and severity of 21 adverse events of antidepressants drugs. For each side effect, a score between 0 (absent) to 3 (severe) is reported. Also, the likelihood of its association with antidepressants is assessed with a yes/no question. Single side-effects scores are summed to obtain a total score (ranging from 0 to 63).
Number of participants with a reduction of at least 50% of the baseline score of the MADRS (responders) | 6 months
  The number of participants with a reduction of at least 50% of the baseline score of the Montgomery-Åsberg Depression Rating Scale (MADRS). The MADRS is a validated rating scale, administered by the clinician, measuring the occurrence and severity of 10 symptomatic dimensions of depression. For each dimension, a score between 0 (normal, no symptoms) to 6 (severely impaired) is reported. Single scores for each dimension are summed to obtain a total score (ranging from 0 to 60).
Efficacy on depressive symptoms as assessed by the MADRS | 6 months
  Mean change scores at MADRS. The MADRS is a validated rating scale, administered by the clinician, measuring the occurrence and severity of 10 symptomatic dimensions of depression. For each dimension, a score between 0 (normal, no symptoms) to 6 (severely impaired) is reported. Single scores for each dimension are summed to obtain a total score (ranging from 0 to 60).
Quality of life as assessed by the EQ-5D | 6 months
  Mean change scores at the EQ-5D. The EQ-5D is a validated rating scale, self-administered, measuring the quality of life according to 5 dimensions. In addition, the overall health status on the day of the interview is measured on a visual analogue scale ranging from 0 (worst possible health status) to 100 (best possible health status). When interpreting the scale, dimensions are to be considered separately and not summed in a total score.
Cognitive performance as assessed by the SBT | 6 months
  Mean change scores at the Short Blessed Scale (SBT). The SBT is a validated rating scale, administered by the clinician, measuring the cognitive performance. The SBT is a screening tool that aids in detecting early cognitive changes associated with dementia disorders. Further testing is warranted if dementia is suspected, the SBT should not be used to diagnose dementia. This is a weighted six-item instrument that evaluates orientation, registration, and attention.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Universitaria Mater Domini, Università Magna Grecia, Catanzaro
  - Sapienza Università di Roma, Dipartimento di Neurologia e Psichiatria, Roma
  - Azienda Ospedaliera Universitaria Verona, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ostuzzi G, Gastaldon C, Barbato A, D'Avanzo B, Tettamanti M, Monti I, Aguglia A, Aguglia E, Alessi MC, Amore M, Bartoli F, Biondi M, Bortolaso P, Callegari C, Carra G, Caruso R, Cavallotti S, Crocamo C, D'Agostino A, De Fazio P, Di Natale C, Giusti L, Grassi L, Martinotti G, Nose M, Papola D, Purgato M, Rodolico A, Roncone R, Tarsitani L, Turrini G, Zanini E, Amaddeo F, Ruggeri M, Barbui C. Tolerability and efficacy of vortioxetine versus SSRIs in elderly with major depression. Study protocol of the VESPA study: a pragmatic, multicentre, open-label, parallel-group, superiority, randomized trial. Trials. 2020 Aug 3;21(1):695. doi: 10.1186/s13063-020-04460-6. PMID 32746941
- [Derived] Bartoli F, Cavaleri D, Riboldi I, Callovini T, Crocamo C, Gastaldon C, Aguglia A, Callegari C, Cavallotti S, Chiappini S, Cruciata M, D'Agostino A, Espa I, Grassi L, Ielmini M, Mammarella S, Martinotti G, Rania M, Rodolico A, Roncone R, Roselli V, Segura-Garcia C, Signorelli MS, Tarsitani L; VESPA Study Group; Ostuzzi G, Carra G. Efficacy and Tolerability of Vortioxetine Versus Selective Serotonin Reuptake Inhibitors for Late-Life Depression: A Post-hoc Analysis of the VESPA Study. Drugs Aging. 2025 Aug;42(8):771-780. doi: 10.1007/s40266-025-01231-3. Epub 2025 Jul 18. PMID 40679716
- [Derived] Ostuzzi G, Gastaldon C, Tettamanti M, Cartabia M, Monti I, Aguglia A, Aguglia E, Bartoli F, Callegari C, Canozzi A, Carbone EA, Carra G, Caruso R, Cavallotti S, Chiappini S, Colasante F, Compri B, D'Agostino A, De Fazio P, de Filippis R, Gari M, Ielmini M, Ingrosso G, Mammarella S, Martinotti G, Rodolico A, Roncone R, Sterzi E, Tarsitani L, Tiberto E, Todini L, Amaddeo F, D'Avanzo B; VESPA Study Group; Barbato A, Barbui C. Tolerability of vortioxetine compared to selective serotonin reuptake inhibitors in older adults with major depressive disorder (VESPA): a randomised, assessor-blinded and statistician-blinded, multicentre, superiority trial. EClinicalMedicine. 2024 Feb 15;69:102491. doi: 10.1016/j.eclinm.2024.102491. eCollection 2024 Mar. PMID 38384338